CLINICAL TRIAL: NCT03337646
Title: A Multi-Center, Open Label, Evaluation of the Effect and Safety of Lisdexamfetamine in Children Aged 6-12 With Attention Deficit Hyperactivity Disorder and Autism Spectrum Disorder
Brief Title: Evaluation of the Effect and Safety of Lisdexamfetamine in Children Aged 6-12 With ADHD and Autism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: JPM van Stralen Medicine Professional (Other)
Collaborators: Shire (Industry)
Responsible Party: Principal Investigator, Dr. Judy van Stralen, Dr. Judy van Stralen, JPM van Stralen Medicine Professional
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RES 16-002
Record Dates: First submitted 2017-11-05; First posted 2017-11-09 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Attention Deficit Hyperactivity Disorder; Autism Spectrum Disorder
Keywords: vyvanse; executive function; safety
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Autism Spectrum Disorder | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Intervention Model Description: Multi-Center Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lisdexamphetamine (Other): All participants will receive Lisdexamfetamine Dimesylate (LDX) at an optimized dose based on protocol
  Interventions: Drug: Lisdexamfetamine Dimesylate

INTERVENTIONS:
Drug: Lisdexamfetamine Dimesylate — Medication to treat ADHD
  Other Names: Vyvanse

SUMMARY:
The purpose of this study is to evaluate the effect and safety of Lisdexamfetamine dimesylate (Vyvanse®) in the treatment of Attention Deficit Hyperactivity Disorder (ADHD) in children and adolescents with ADHD and comorbid Autism Spectrum Disorder (ASD). This would be a novel study as there is no known safety or efficacy data for amphetamine based medications in this population. In addition, although health related quality of life and executive function are known to improve with the treatment of lisdexamfetamine dimesylate in the ADHD population (Banaschewski 2013; Findling 2009; Turgay 2010), it has not been shown in the co-morbid ADHD and ASD population. ADHD is the most common pediatric neurobiological condition affecting approximately five percent of the pediatric population (Feldman 2009). ASD is being increasingly recognized as affecting a substantial amount of the pediatric population, with recent prevalence data showing 1 in 68 affected (Baio, 2014). Prior to the introduction of DSM-5 (APA, 2013), exclusion criteria precluded the diagnosis of ADHD when ASD was present. Studies have shown that 41%-71% of children with ASD also meet criteria for ADHD (Goldstein 2004, Sturm 2004,Yoshida 2004, Gadow 2006). This means that up to 1% of the population may have co-morbid ADHD and ASD. With the official recognition of this comorbidity, treatment of comorbid ADHD when ASD is also present has been increasingly recognized as an important strategy in improving executive functioning and quality of life in those affected. Studies have indicated that some of the medications commonly used to treat ADHD, are effective and safe when used in comorbid ADHD and ASD. At this time, there have been well designed studies demonstrating safety and efficacy for methylphenidate (Ghuman et al. 2009; Handen et al. 2000; Quintana et al. 1995; RUPP 2005), guanfacine XR (Posey 2004; Scahill 2015), and atomoxetine (Arnold 2006; Harfterkamp 2012).

DETAILED DESCRIPTION:
ADHD is the most common pediatric neurobiological condition affecting approximately five percent of the pediatric population (Faraone, Stephen V., Sergeant, J. et al. 2003; Feldman & Belanger 2009). ASD is being increasingly recognized as affecting a substantial amount of the pediatric population, with recent prevalence data showing 1 in 68 affected (U.S. Department of Health and Human Services 2010). Prior to the introduction of DSM-5, exclusion criteria precluded the diagnosis for ADHD when ASD was present (American Psychiatric Association 2013). Studies have shown that 41%-71% of children with ASD also meet criteria for ADHD, meaning up to 1% of the population may have comorbid ADHD and ASD (Goldstein & Schewbach 2004).

With the official recognition of comorbidity, treatment of comorbid ADHD when ASD is also present has been increasingly recognized as an important strategy in decreasing ADHD symptoms, and improving executive functioning and quality of life of those affected. Studies have indicated that some of the medications (methylphenidate, guanfacine XR and atomoxetine) commonly used to treat ADHD are effective and safe when used in comorbid ADHD and ASD (Ornstein & Kollins 2012; Ghuman et al. 2009; Handen et al. 2000; Quintana et al. 1995; Posey et al. 2004; Scahill et al. 2015; M. et al. 2012). While amphetamine class compounds are amongst the first line of treatment in ADHD, the lack of studies in this population has discouraged their use in subjects with comorbid ADHD and ASD.

The lack of safety and efficacy data is problematic as it limits therapeutic options for the population of subjects with ADHD and ASD. Amphetamines and methylphenidate medications are equally considered first line treatment options for ADHD (CADDRA 2011). Some subjects may preferentially respond to one group of medications over another, therefore it is important to have clear safety and efficacy data for both therapeutic options.

A retrospective chart review of this population indicates that treatment is started with methylphenidate versus combined amphetamine/dextroamfetamine at a ratio of 2.78:1 (Stigler et al. 2004). Due to the availability of evidence of efficacy in this comorbid population, clinicians may choose to skip to what is considered a second line medication for ADHD symptomatology rather than using LDX (or another amphetamine-based ADHD medication such as dexedrine or Adderall XR) that may have a larger effect size for treating these symptoms.

LDX has been shown to be an effective treatment for ADHD in subjects 6 and above. With long lasting effectiveness shown to last up to 14 hours, it could potentially improve ADHD symptoms and overall quality of life for children and adolescents with ADHD and ASD in home, school and after-school functioning.

The purpose of this study is to evaluate the safety and efficacy of LDX in treating ADHD when ASD is co-morbid.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject aged 6-12 years at the time of consent/assent.
2. Subjects parent(s) or legally authorized representative (LAR) must provide signature of informed consent, and there must be documentation of assent (if applicable) by the subject in accordance with the International Council on Harmonisation (ICH) Good Clinical Practice (GCP) Guideline E6 (1996), any updates or revisions, and applicable regulations, before completing any study related procedures.
3. Subject and parent(s)/LAR are willing and able to comply with all of the requirements defined in the protocol.
4. Subject meets Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-V) criteria for a diagnosis of ADHD combined presentation, inattentive presentation or hyperactive/impulsive presentation based on history and a minimum ADHD-RS score of 32 and a minimum CGI-S of 4 at baseline.
5. Subject meets DSM-V criteria for a diagnosis of ASD-level 1 based on history and Autism Diagnostic Observation Scale (ADOS-2).
6. Subject has an SRS-2 total score of ≥ 70.
7. Subject has a Clinical Global Impressions - Severity of Illness (CGI-S) score ≥ 4 at the baseline visit (visit 2)
8. Subject has a blood pressure measurement within 95th percentile for age, and sex (Appendix 1,1.1,2 & 2.2). Subject and parent/legally authorized representative (LAR) are willing, able and likely to comply with the study procedures and restrictions within the protocol.

Exclusion Criteria:

1. Subject has any condition that, in the opinion of the investigator, represent an inappropriate risk to the subject or may confound the interpretation of the study.
2. Subject has a known history or presence of structural cardiac abnormalities, cardiovascular or cerebrovascular disease, serious heart rhythm abnormalities, syncope, tachycardia, cardiac conduction problems (such as clinically significant heart block or QT interval prolongation), exercise-related cardiac events including syncope and pre-syncope or clinically significant bradycardia.
3. Subject has a known history of symptomatic cardiovascular disease, unexplained syncope, exertional chest pain, advanced arteriosclerosis, structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormalities, coronary artery disease or other serious cardiac problems placing them at increased vulnerability to sympathomimetic effects of a stimulant drug.
4. Subject has a history of seizure disorder (other than a single childhood febrile seizure occurring before the age of 3 years).
5. Subject has glaucoma.
6. Subject is currently using prohibited medication.
7. Subject has a known or suspected allergy, hypersensitivity, or clinically significant intolerance to LDX.
8. Subject has taken another investigational product within 30 day prior to baseline.
9. Subject has initiated behavioural therapy within 1 month of the baseline visit (visit 0). Subject may not initiate behavioural therapy during the study.
10. Subject is female and is pregnant or currently lactating.
11. Subject is currently considered a suicide risk in the opinion of the investigator, has previously made a suicide attempt, or has a prior history of or is currently demonstrating active suicide ideation. Subjects with intermittent passive suicidal ideation are not necessarily excluded based on the assessment of the investigator.
12. History of failure to respond to an adequate trial of an amphetamine based medication.
13. Subject is currently abusing an illicit substance or lives with someone known to currently abuse stimulants or cocaine..
14. Subject has a known renal or hepatic insufficiency.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
ADHD Symptoms | 12 weeks
  Physician rated scale ADHD IV-RS each item is scaled 1 to 3 with a total between 0 and 54

SECONDARY OUTCOMES:
Health Related Quality of Life | 12 weeks
  Parent completed rating scale called Child Health and Illness Profile- Child Edition: Parent Report Form ( CHIP-CE-PRF) . This is a generic child health status questionnaire that comprehensively describes all aspects of child health that can be influenced by the health care and school systems. It includes subdomains of satisfaction, discomfort, resilience, risk avoidance, achievement, and disorders. The domains and subdomains were conceptually derived and generally supported by factor analysis. The majority of items assess frequency of behaviors or experiences. Most items use a five-point response format. When a recall period is used, it is typically the past 4 weeks. Scale scores are obtained by computing the average of the individual item responses, whether scoring the domain or subdomain (in the PRF). The scale scores are standardized with a mean of 50 and standard deviation of 10. Higher scores indicate better health.
Executive Function | 12 weeks
  The BRIEF-P is a 90 item parent completed questionnaire with a global executive composite score (GEC). GEC is reported as a t-score and a t-score of less than 65 is within normal limits
Severity of illness | 12 weeks
  The severity of illness using the Clinical Global Impression-severity of illness, a 7 point scale which is physician rated
Improvement of Subjects | 12 weeks
  The severity of illness using the Clinical Global Impression-improvement of illness, a 7 point scale which is physician rated To evaluate the change in functional impairment in subjects. A score of 1 indicates very much improved while a score of 7 indicates very much worse
Safety-Adverse events | 12 weeks
  Adverse events are recorded at every visit
Safety - suicidality | 12 weeks
  Using the Columbia-Suicide Severity Rating Scale the incidence of suicidal thoughts and actions are recorded. The C-SSRS (Posner et al. 2011; Posner et al. 2010) is a semi-structured interview that captures the occurrence, severity, and frequency of suicide-related thoughts and behaviours during the assessment period. The interview includes definitions and suggested questions to solicit the type of information needed to determine if a suicide-related thought or behaviour has occurred.

CONTACTS AND LOCATIONS:
Overall Officials: Judy van Stralen, MD, Principal Investigator — Center for Pediatric Excellence
Locations (1):
- Center for Pediatric Excellence, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] First MB. Diagnostic and statistical manual of mental disorders, 5th edition, and clinical utility. J Nerv Ment Dis. 2013 Sep;201(9):727-9. doi: 10.1097/NMD.0b013e3182a2168a. No abstract available. PMID 23995026
- [Background] Arnsten AF. Modulation of prefrontal cortical-striatal circuits: relevance to therapeutic treatments for Tourette syndrome and attention-deficit hyperactivity disorder. Adv Neurol. 2001;85:333-41. No abstract available. PMID 11530441
- [Background] Bhutta AT, Cleves MA, Casey PH, Cradock MM, Anand KJ. Cognitive and behavioral outcomes of school-aged children who were born preterm: a meta-analysis. JAMA. 2002 Aug 14;288(6):728-37. doi: 10.1001/jama.288.6.728. PMID 12169077
- [Background] Biederman J, Krishnan S, Zhang Y, McGough JJ, Findling RL. Efficacy and tolerability of lisdexamfetamine dimesylate (NRP-104) in children with attention-deficit/hyperactivity disorder: a phase III, multicenter, randomized, double-blind, forced-dose, parallel-group study. Clin Ther. 2007 Mar;29(3):450-63. doi: 10.1016/s0149-2918(07)80083-x. PMID 17577466
- [Background] Bolte S, Willfors C, Berggren S, Norberg J, Poltrago L, Mevel K, Coco C, Fransson P, Borg J, Sitnikov R, Toro R, Tammimies K, Anderlid BM, Nordgren A, Falk A, Meyer U, Kere J, Landen M, Dalman C, Ronald A, Anckarsater H, Lichtenstein P. The Roots of Autism and ADHD Twin Study in Sweden (RATSS). Twin Res Hum Genet. 2014 Jun;17(3):164-76. doi: 10.1017/thg.2014.12. Epub 2014 Apr 15. PMID 24735654
- [Background] Brown K. Neuroscience. New attention to ADHD genes. Science. 2003 Jul 11;301(5630):160-1. doi: 10.1126/science.301.5630.160. No abstract available. PMID 12855786
- [Background] Bruni, T., 2014. Test Review: Social Responsiveness Scale-Second Edition. (SRS-2).
- [Background] Coghill DR, Caballero B, Sorooshian S, Civil R. A systematic review of the safety of lisdexamfetamine dimesylate. CNS Drugs. 2014 Jun;28(6):497-511. doi: 10.1007/s40263-014-0166-2. PMID 24788672
- [Background] Department of Health, E. and W., 1976. Clinical Global Impression (CGI). In Guy W. ED. ECEDEU Assessment Manual for pyschopharmacology.
- [Background] DuPaul, G. et al., 1998. ADHD Rating Scale IV: Checklists, Norms and Clinical Interpretation. In New York, NY: Guilford Press.
- [Background] Efron D, Jarman F, Barker M. Side effects of methylphenidate and dexamphetamine in children with attention deficit hyperactivity disorder: a double-blind, crossover trial. Pediatrics. 1997 Oct;100(4):662-6. doi: 10.1542/peds.100.4.662. PMID 9310521
- [Background] Faraone SV, Sergeant J, Gillberg C, Biederman J. The worldwide prevalence of ADHD: is it an American condition? World Psychiatry. 2003 Jun;2(2):104-13. PMID 16946911
- [Background] Faraone SV. Lisdexamfetamine dimesylate: the first long-acting prodrug stimulant treatment for attention deficit/hyperactivity disorder. Expert Opin Pharmacother. 2008 Jun;9(9):1565-74. doi: 10.1517/14656566.9.9.1565. PMID 18518785
- [Background] Feldman M, Belanger S. Extended-release medications for children and adolescents with attention-deficit hyperactivity disorder. Paediatr Child Health. 2009 Nov;14(9):593-602. doi: 10.1093/pch/14.9.593. PMID 21037836
- [Background] Ghuman JK, Aman MG, Lecavalier L, Riddle MA, Gelenberg A, Wright R, Rice S, Ghuman HS, Fort C. Randomized, placebo-controlled, crossover study of methylphenidate for attention-deficit/hyperactivity disorder symptoms in preschoolers with developmental disorders. J Child Adolesc Psychopharmacol. 2009 Aug;19(4):329-39. doi: 10.1089/cap.2008.0137. PMID 19702485
- [Background] Gioia, G. et al., 2000. Behaviour Rating Inventory of Executive Function (BRIEF): Professional Manual,
- [Background] Goldstein S, Schwebach AJ. The comorbidity of Pervasive Developmental Disorder and Attention Deficit Hyperactivity Disorder: results of a retrospective chart review. J Autism Dev Disord. 2004 Jun;34(3):329-39. doi: 10.1023/b:jadd.0000029554.46570.68. PMID 15264500
- [Background] Handen BL, Johnson CR, Lubetsky M. Efficacy of methylphenidate among children with autism and symptoms of attention-deficit hyperactivity disorder. J Autism Dev Disord. 2000 Jun;30(3):245-55. doi: 10.1023/a:1005548619694. PMID 11055460
- [Background] Hardman, J., Limbird, L. & Gilman, A., 2001. Goodman & Gillman's The Pharmacological Basis of Therapeutics, 10th edition,
- [Background] Hazlett HC, Poe M, Gerig G, Smith RG, Provenzale J, Ross A, Gilmore J, Piven J. Magnetic resonance imaging and head circumference study of brain size in autism: birth through age 2 years. Arch Gen Psychiatry. 2005 Dec;62(12):1366-76. doi: 10.1001/archpsyc.62.12.1366. PMID 16330725
- [Background] Heal DJ, Smith SL, Gosden J, Nutt DJ. Amphetamine, past and present--a pharmacological and clinical perspective. J Psychopharmacol. 2013 Jun;27(6):479-96. doi: 10.1177/0269881113482532. Epub 2013 Mar 28. PMID 23539642
- [Background] Kratochvil CJ, Vaughan BS, Harrington MJ, Burke WJ. Atomoxetine: a selective noradrenaline reuptake inhibitor for the treatment of attention-deficit/hyperactivity disorder. Expert Opin Pharmacother. 2003 Jul;4(7):1165-74. doi: 10.1517/14656566.4.7.1165. PMID 12831341
- [Background] Kahn RS, Khoury J, Nichols WC, Lanphear BP. Role of dopamine transporter genotype and maternal prenatal smoking in childhood hyperactive-impulsive, inattentive, and oppositional behaviors. J Pediatr. 2003 Jul;143(1):104-10. doi: 10.1016/S0022-3476(03)00208-7. PMID 12915833
- [Background] Leitner Y. The co-occurrence of autism and attention deficit hyperactivity disorder in children - what do we know? Front Hum Neurosci. 2014 Apr 29;8:268. doi: 10.3389/fnhum.2014.00268. eCollection 2014. PMID 24808851
- [Background] Lewin AH, Miller GM, Gilmour B. Trace amine-associated receptor 1 is a stereoselective binding site for compounds in the amphetamine class. Bioorg Med Chem. 2011 Dec 1;19(23):7044-8. doi: 10.1016/j.bmc.2011.10.007. Epub 2011 Oct 13. PMID 22037049
- [Background] Lord C, Cook EH, Leventhal BL, Amaral DG. Autism spectrum disorders. Neuron. 2000 Nov;28(2):355-63. doi: 10.1016/s0896-6273(00)00115-x. No abstract available. PMID 11144346
- [Background] Harfterkamp M, van de Loo-Neus G, Minderaa RB, van der Gaag RJ, Escobar R, Schacht A, Pamulapati S, Buitelaar JK, Hoekstra PJ. A randomized double-blind study of atomoxetine versus placebo for attention-deficit/hyperactivity disorder symptoms in children with autism spectrum disorder. J Am Acad Child Adolesc Psychiatry. 2012 Jul;51(7):733-41. doi: 10.1016/j.jaac.2012.04.011. Epub 2012 May 25. PMID 22721596
- [Background] Davis NO, Kollins SH. Treatment for co-occurring attention deficit/hyperactivity disorder and autism spectrum disorder. Neurotherapeutics. 2012 Jul;9(3):518-30. doi: 10.1007/s13311-012-0126-9. PMID 22678458
- [Background] Posey DJ, Puntney JI, Sasher TM, Kem DL, McDougle CJ. Guanfacine treatment of hyperactivity and inattention in pervasive developmental disorders: a retrospective analysis of 80 cases. J Child Adolesc Psychopharmacol. 2004 Summer;14(2):233-41. doi: 10.1089/1044546041649084. PMID 15319020
- [Background] Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oquendo MA, Currier GW, Melvin GA, Greenhill L, Shen S, Mann JJ. The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry. 2011 Dec;168(12):1266-77. doi: 10.1176/appi.ajp.2011.10111704. PMID 22193671
- [Background] Quintana H, Birmaher B, Stedge D, Lennon S, Freed J, Bridge J, Greenhill L. Use of methylphenidate in the treatment of children with autistic disorder. J Autism Dev Disord. 1995 Jun;25(3):283-94. doi: 10.1007/BF02179289. PMID 7559293
- [Background] Scahill L, McCracken JT, King BH, Rockhill C, Shah B, Politte L, Sanders R, Minjarez M, Cowen J, Mullett J, Page C, Ward D, Deng Y, Loo S, Dziura J, McDougle CJ; Research Units on Pediatric Psychopharmacology Autism Network. Extended-Release Guanfacine for Hyperactivity in Children With Autism Spectrum Disorder. Am J Psychiatry. 2015 Dec;172(12):1197-206. doi: 10.1176/appi.ajp.2015.15010055. Epub 2015 Aug 28. PMID 26315981
- [Background] Stigler KA, Desmond LA, Posey DJ, Wiegand RE, McDougle CJ. A naturalistic retrospective analysis of psychostimulants in pervasive developmental disorders. J Child Adolesc Psychopharmacol. 2004 Spring;14(1):49-56. doi: 10.1089/104454604773840481. PMID 15142391
- [Background] Thomas R, Sanders S, Doust J, Beller E, Glasziou P. Prevalence of attention-deficit/hyperactivity disorder: a systematic review and meta-analysis. Pediatrics. 2015 Apr;135(4):e994-1001. doi: 10.1542/peds.2014-3482. Epub 2015 Mar 2. PMID 25733754
- [Background] Thompson T, Lloyd A, Joseph A, Weiss M. The Weiss Functional Impairment Rating Scale-Parent Form for assessing ADHD: evaluating diagnostic accuracy and determining optimal thresholds using ROC analysis. Qual Life Res. 2017 Jul;26(7):1879-1885. doi: 10.1007/s11136-017-1514-8. Epub 2017 Feb 20. PMID 28220338
- [Background] U.S. Department of Health and Human Services, 2010. Prevalence of autism spectrum disorder among children aged 8 years - autism and developmental disabilities
- See also: CADDRA, 2011. Canadian ADHD Practice Guidelines, — http://www.caddra.ca
- See also: Riley, A.W. et al., 2004. The Parent Report Form of the CHIP Child Edition. Medical Care, 42(3), pp.210-220. . — https://pubmed.ncbi.nlm.nih.gov/15076820/